CLINICAL TRIAL: NCT03706274
Title: A Phase 1, Open-Label, Dose-Ranging Study of the PD-1 Probody Therapeutic CX-188 in Adults With Recurrent or Metastatic Solid Tumors
Brief Title: PROCLAIM-CX-188: A Trial to Find Safe and Active Doses of an Investigational Drug CX-188 for Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: CytomX Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMX-M-188-001
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CX-188 Escalation (Experimental)
  Interventions: Drug: CX-188
- CX-188 Alternative Dosing Schedule (Experimental)
  Interventions: Drug: CX-188

INTERVENTIONS:
Drug: CX-188 — CX-188

SUMMARY:
The purpose of this first-in-human study of CX-188 is to characterize the safety, tolerability, pharmacokinetics (PK), and antitumor activity of CX-188 in adult subjects with metastatic or advanced unresectable solid tumors that progressed on standard therapy: PROCLAIM: PRObody Clinical Assessment in Man CX-188 clinical trial 001

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed diagnosis of metastatic or advanced unresectable solid tumors that progressed on standard therapy
2. agreement to provide mandatory archival tumor or fresh biopsy before they can be considered for inclusion in the study 3. At least 18 years old

Exclusion Criteria:

1. Prior therapy with a chimeric antigen receptor (CAR) T-cell containing regimen.
2. History of severe allergic or anaphylactic reactions to human monoclonal antibody therapy or known hypersensitivity to any Probody therapeutic
3. Human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)-related illness, chronic hepatitis B or C
4. History of or current active autoimmune diseases
5. History of syndrome or medical condition(s) that requires systemic steroids (> 10 mg daily prednisone equivalents) or immunosuppressive medications
6. History of allogeneic tissue/solid organ transplant, prior stem cell or bone marrow transplant
7. Chemotherapy, biochemotherapy, radiation or immunotherapy or any investigational treatment within 30 days prior to receiving any study drug
8. Major surgery (requiring general anesthesia) within 3 months or minor surgery (excluding biopsies conducted with local/topical anesthesia) or gamma knife treatment within 14 days (with adequate healing) of administration of any study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The number of subjects experiencing a dose-limiting toxicity at various dose levels when given CX-188 as a monotherapy | 21 days

SECONDARY OUTCOMES:
The percentage of subjects experiencing anti-cancer activity (ORR) at various dose levels when given CX-188 as monotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yifah Yaron, MD, Study Director — CytomX Therapeutics
Locations (1):
- Virginia Cancer Specialists, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No